CLINICAL TRIAL: NCT00718393
Title: Compassionate Use of Ceftriaxone in Patients With ALS
Brief Title: Compassionate Use of Ceftriaxone in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Type: Observational
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-16964
Record Dates: First submitted 2008-07-14; First posted 2008-07-18 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.

SUMMARY:
Amyotrophic lateral sclerosis is a uniformly progressive and fatal neurodegenerative disorder for which there is no known cure. In a novel attempt to widen the search for potential therapeutic agents, a NINDS- led cooperative group performed an in-vitro screening program of 1040 FDA approved drugs in over 28 assays relevant to various neurodegenerative disorders. Several cephalosporins showed hits in ALS relevant assays. Efficacy was noted in models suggesting increased expression of the astrocytic glutamate transporter, EAAT2, as well as models of superoxide dismutase mediated toxicity. Ceftriaxone is a third generation cephalosporin with good CNS penetration, a long half-life, and was effective in both types of ALS assays. Ceftriaxone has calcium binding activity, antioxidant properties, and rescues motor neurons in culture from chronic glutamate toxicity. Since completion of the original NINDS screen, Ceftriaxone has been shown to increase by three fold EAAT2 activity in rodent brains, due to ceftriaxone's ability to increase EAAT2 promotor activation This program is for the use of ceftriaxone in ALS for compassionate care. Currently ceftriaxone is approved by the U.S. Food and Drug Administration (FDA) for treating bacterial infections but not for treating ALS. However, there is an ongoing phase I study -by NEALS Consortium and the National Institute of Health- with three cohorts -a placebo group and two groups receiving either 2 or 4 grams of ceftriaxone daily-. Unfortunately there are only a limited number of patients being enrolled and the next phase of the project will not be undertaken until next year. At this point there are ALS patients unable to participate in this Phase I trial and unlikely to be alive when the next phase of study begins. Some of these patients want to receive the drug and are willing to pay for the drug and nursing care. We are therefore requesting a compassionate use protocol for these patients who request the medication and are willing to pay for the drug and nursing care to administer it. Dr. Terry Heiman-Patterson will supervise the administration and safety monitoring including labs for renal and hepatic function as well as IV site inspection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or probable ALS by the El Escorial Criteria
* Participants must be medically able to undergo the study procedures
* Subjects must have a registered nurse who can administer the drug daily and also inspect the IV site
* Not Pregnant
* Willing to pay for the cost of drug, administration, and safety testing
* Able to give informed consent

Exclusion Criteria:

* Patients who are not diagnosed with ALS by a physician
* Patients unable to give informed consent
* Patients who have a history of sensitivity to cephalosporin or penicillin antibiotics (such as Ancef, Keflex, Ceclor, Ceftin, Lorabid, Suprax, or Fortaz).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS clinic patients at MDA/ALS Center of Hope.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

IPD SHARING:
Plan to Share IPD: No